CLINICAL TRIAL: NCT07215299
Title: Temporal Interference Methods for Non-invasive Deep Brain Stimulation
Brief Title: Temporal Interference Methods for Non-invasive Deep Brain Stimulation, Study 1.1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joshua Brown, PHD, Professor of Pyschological and Brain Science, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 26941, Study 1.1; 1R21MH140210-01 (NIH)
Record Dates: First submitted 2025-09-29; First posted 2025-10-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers
Keywords: Temporal Interference; fMRI; BOLD Signal; Cognitive Control; Dorsal Anterior Cingulate Cortex; Non-invasive deep brain stimulation; Neurostimulation

STUDY DESIGN:
Intervention Model Description: This study uses a within-subject crossover design. Participants receive both active temporal interference (TI) stimulation and sham stimulation, in both "on" and "off" conditions during fMRI scanning. The order of active vs. sham stimulation and the order of on vs off conditions is counterbalanced across participants. Beat frequency, electrode placement, and behavioral paradigm vary by sub-study (e.g., reward-related tasks targeting the nucleus accumbens, cognitive control and decision-making tasks targeting the dorsal anterior cingulate cortex). For Study 1.1, a 20Hz beat frequency will be evaluated for its effect on the nucleus accumbens.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- NAcc TI Active, then NAcc TI Sham, then NAcc No-TI Active, then NAcc No-TI Sham (Active Comparator): Participants in this Arm receive temporal interference (TI) electrical stimulation with two pairs of carbon fiber electrodes in this order: NAcc TI Active, then NAcc TI Sham, then NAcc No-TI Active, then NAcc No-TI Sham.
  Interventions: Device: Temporal Interference (TI) Electrical Stimulation - NAcc TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc TI Sham; Device: Temporal Interference (TI) Electrical Stimulation - NAcc No-TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc No-TI Sham
- NAcc No-TI Active, then NAcc No-TI Sham, then NAcc TI Active, then NAcc TI Sham (Active Comparator): Participants in this Arm receive temporal interference (TI) electrical stimulation with two pairs of carbon fiber electrodes in this order: NAcc No-TI Active, then NAcc No-TI Sham, then NAcc TI Active, then NAcc TI Sham.
  Interventions: Device: Temporal Interference (TI) Electrical Stimulation - NAcc TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc TI Sham; Device: Temporal Interference (TI) Electrical Stimulation - NAcc No-TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc No-TI Sham
- NAcc TI Sham, then NAcc TI Active, then NAcc No-TI Sham, then NAcc No-TI Active (Active Comparator): Participants in this Arm receive temporal interference (TI) electrical stimulation with two pairs of carbon fiber electrodes in this order: NAcc TI Sham, then NAcc TI Active, then NAcc No-TI Sham, then NAcc No-TI Active.
  Interventions: Device: Temporal Interference (TI) Electrical Stimulation - NAcc TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc TI Sham; Device: Temporal Interference (TI) Electrical Stimulation - NAcc No-TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc No-TI Sham
- NAcc No-TI Sham, then NAcc No-TI Active, then NAcc TI Sham, then NAcc TI Active (Active Comparator): Participants in this Arm receive temporal interference (TI) electrical stimulation with two pairs of carbon fiber electrodes in this order: NAcc No-TI Sham, then NAcc No-TI Active, then NAcc TI Sham, then NAcc TI Active.
  Interventions: Device: Temporal Interference (TI) Electrical Stimulation - NAcc TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc TI Sham; Device: Temporal Interference (TI) Electrical Stimulation - NAcc No-TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc No-TI Sham

INTERVENTIONS:
Device: Temporal Interference (TI) Electrical Stimulation - NAcc TI Active — Non-invasive electrical brain stimulation delivered through two sets of scalp electrodes using alternating current frequencies (e.g., 2000 Hz and 2020 Hz) at up to 2 mA per electrode. This stimulation creates a beat frequency interference pattern (e.g., 20 Hz) that focally stimulates deep brain regions without activating overlying cortex.
  For the NAcc TI Active condition, 2000Hz will be administered in one channel and 2020Hz in the other. These frequencies will be administered in 2 minutes on/2 minutes off cycles with a 30 second ramp up and ramp down beginning at the start of each 2 minute period.
  Other Names: TI Electrical Neurostimulation; TI Neurostimulation
Device: Temporal Interference (TI) Electrical Stimulation - NAcc TI Sham — Non-invasive electrical brain stimulation delivered through two sets of scalp electrodes using alternating current frequencies (e.g., 2000 Hz and 2020 Hz) at up to 2 mA per electrode. This stimulation creates a beat frequency interference pattern (e.g., 20 Hz) that focally stimulates deep brain regions without activating overlying cortex.
  For the NAcc TI Sham condition, 2000Hz will be administered in one channel and 2020Hz in the other. These frequencies will be administered in 2 minutes on/2 minutes off cycles, however, instead of the 30 second ramp up and ramp down at the beginning of each 2 minute period (as seen in the Active TI condition), the stimulation in the NAcc TI Sham condition will immediately ramp down as soon as it reaches 2mA after ramp up.
  Other Names: TI Electrical Neurostimulation; TI Neurostimulation
Device: Temporal Interference (TI) Electrical Stimulation - NAcc No-TI Active — Non-invasive electrical brain stimulation delivered through two sets of scalp electrodes using the same current frequencies at up to 2 mA per electrode.
  For the NAcc No-TI Active condition, 2000Hz will be administered in both channels. These frequencies will be administered in 2 minutes on/2 minutes off cycles with a 30 second ramp up and ramp down beginning at the start of each 2 minute period.
  Other Names: TI Electrical Neurostimulation; TI Neurostimulation
Device: Temporal Interference (TI) Electrical Stimulation - NAcc No-TI Sham — Non-invasive electrical brain stimulation delivered through two sets of scalp electrodes using the same current frequencies at up to 2 mA per electrode.
  For the NAcc No-TI Sham condition, 2000Hz will be administered in both channels. These frequencies will be administered in 2 minutes on/2 minutes off cycles, however, instead of the 30 second ramp up and ramp down at the beginning of each 2 minute period (as seen in the NAcc No-TI Active condition), the stimulation in the NAcc No-TI Sham condition will immediately ramp down as soon as it reaches 2mA after ramp up.
  Other Names: TI Electrical Neurostimulation; TI Neurostimulation

SUMMARY:
In its totality, this grant aims to develop a line of research using temporal interference (TI) electrical neurostimulation technology to understand the causal role of deep brain structures in cognition. In the short term, the investigators aim to validate and characterize the effects of TI on brain activity as measured by fMRI and demonstrate its ability to focally stimulate deep brain regions without affecting overlying cortex. In the longer term, investigators aim to use these data to resolve longstanding debates about the function of deeper brain regions and lay the foundation for future clinical applications of TI for treating addiction, Obsessive-Compulsive Disorder (OCD), Parkinson's disease, and other disorders involving deep brain dysfunction. The grant supports 2 distinct aims, each of which will be evaluated through a series of independent studies.

DETAILED DESCRIPTION:
Through the grant's duration, the investigators hypothesize that temporal interference (TI) electrical neurostimulation will be well tolerated and effective at focally manipulating deep brain activity as measured by functional MRI (fMRI) BOLD signals. The investigators will investigate whether TI stimulation can increase BOLD activity in targeted deep brain regions including the nucleus accumbens (NAcc) and dorsal anterior cingulate cortex (dACC), and whether this stimulation can influence cognitive functions controlled by these regions. TI works by applying alternating currents of slightly different frequencies through multiple electrode pairs, creating an interference pattern that can stimulate deep brain regions without significantly affecting superficial cortical areas. This method is similar to traditional transcranial direct current stimulation (tDCS), however TI can stimulate deeper brain structures that tDCS cannot reach effectively. The study is broken up into two main aims with multiple sub-studies. In Aim 1, the investigators will characterize the effects of TI on fMRI BOLD signals, test different beat frequencies, and compare TI effects in the nucleus accumbens versus dorsal anterior cingulate cortex. In Aim 2, the investigators will apply TI to the dorsal anterior cingulate cortex to test causal theories about its role in cognitive control, conflict monitoring, risk avoidance, and foraging behavior using established cognitive tasks while subjects undergo fMRI scanning.

Study 1.1 (Aim 1, Study 1) will test the ability to focally activate the nucleus accumbens without activating the overlying cortex, and also its effects on functional connectivity. Healthy subjects (n=30) will present for a single study visit during which they will be placed in the fMRI scanner and administered a temporal interference protocol. Specifically, subjects will have two pairs of carbon fiber electrodes attached to the scalp with conductive gel. They will receive one 8-minute block of stimulation at 2mA per electrode pair. The stimulation sequence will be 2 minutes on, 2 minutes off, 2 minutes on, and 2 minutes off with 30 second ramp up and ramp down beginning at the start of each 2-minute period. The first block will apply active TI stimulation with 2000Hz in one channel and 2020Hz in the other channel. The second block will be a sham TI stimulation, identical to the first block but with the "on" condition immediately ramping down as soon as it reaches 2mA after ramp up. The third and fourth blocks will be identical to the first and second blocks, except that both electrode pairs will stimulate at 2000Hz, resulting in a "NO-TI active" and "NO-TI sham" conditions. The order of blocks, and whether the "on" or "off" condition occurs first within a block, will be counterbalanced across subjects.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 50
* Must have at least a 6th grade education
* Ability to speak and read English for all phases

Exclusion Criteria:

* Currently taking psychotropic medications for ADHD, other mental illness, or medications for cancer
* History of epilepsy or seizure disorders
* History of migraines or other neurological syndromes
* History of AIDS (due to potential cognitive deficits)
* History of head trauma or cognitive impairments
* Personal experiences consistent with symptoms of psychosis (e.g., hallucinations, delusions of control or special powers)
* History of skull defects (e.g., holes bored into the skull or known cranial fissures)
* Metal implants in the head or under the scalp
* Does not meet fMRI safety screening criteria (e.g., metal implants in the body, permanent jewelry, tattoos on the head or neck)
* Uses an intrauterine device (IUD) for birth control and cannot provide documentation to verify MRI safety
* Pregnancy (self-reported; no pregnancy test administered)
* Weight over 440 lbs (scanner weight limit)
* Presence of pacemakers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Change in brain activity in the nucleus accumbens during active versus sham stimulation | During fMRI scan on study day (approximately 60 minutes)
  Brain activity in the nucleus accumbens will be measured using functional magnetic resonance imaging (fMRI) during active temporal interference (TI) brain stimulation compared to sham (placebo) stimulation. Activity will be reported as the percent change in blood-oxygen-level-dependent (BOLD) signal, which reflects changes in brain activity. Higher BOLD values indicate stronger brain activation.

SECONDARY OUTCOMES:
Change in brain activity in the nucleus accumbens during no-TI active versus no-TI sham high-frequency stimulation | During fMRI scan on study day (approximately 60 minutes)
  Brain activity will be measured using fMRI when both electrode pairs deliver the same frequency (no-TI control). The percent change in BOLD signal during active versus sham high-frequency stimulation will be compared to determine whether high-frequency stimulation alone changes brain activity.
Change in brain activity in the nucleus accumbens during active TI stimulation versus active no-TI stimulation | During fMRI scan on study day (approximately 60 minutes)
  Brain activity in the nucleus accumbens will be compared between active TI stimulation and active high-frequency (no-TI) stimulation. This comparison will show whether TI stimulation produces greater activation than high-frequency stimulation alone. Activity will be reported as the percent change in blood-oxygen-level-dependent (BOLD) signal, which reflects changes in brain activity. Higher BOLD values indicate stronger brain activation.
Change in brain connectivity between the nucleus accumbens and other brain regions during stimulation | During fMRI scan on study day (approximately 60 minutes)
  Functional connectivity between the nucleus accumbens and other brain regions will be measured using fMRI-based analyses during active versus sham TI stimulation. Higher correlation values indicate stronger communication between brain regions. Activity will be reported as the percent change in blood-oxygen-level-dependent (BOLD) signal, which reflects changes in brain activity. Higher BOLD values indicate stronger brain activation. The test statistic will be the whole-brain interaction term of seed region BOLD activity multiplied by the condition of active vs. sham TI, more commonly known as a psycho-physiological interaction test.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua W Brown, PhD, Principal Investigator — Indiana University, Bloomington
Locations (1):
- Indiana University Bloomington, Imaging Research Facility, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Violante IR, Alania K, Cassara AM, Neufeld E, Acerbo E, Carron R, Williamson A, Kurtin DL, Rhodes E, Hampshire A, Kuster N, Boyden ES, Pascual-Leone A, Grossman N. Non-invasive temporal interference electrical stimulation of the human hippocampus. Nat Neurosci. 2023 Nov;26(11):1994-2004. doi: 10.1038/s41593-023-01456-8. Epub 2023 Oct 19. Erratum In: Nat Neurosci. 2023 Dec;26(12):2252. doi: 10.1038/s41593-023-01517-y. PMID 37857775
- [Background] Modak P, Fine J, Colon B, Need E, Cheng H, Hulvershorn L, Finn P, Brown JW. Temporal interference electrical neurostimulation at 20 Hz beat frequency leads to increased fMRI BOLD activation in orbitofrontal cortex in humans. Brain Stimul. 2024 Jul-Aug;17(4):867-875. doi: 10.1016/j.brs.2024.07.014. Epub 2024 Jul 24. PMID 39059712
- [Background] Grossman N, Bono D, Dedic N, Kodandaramaiah SB, Rudenko A, Suk HJ, Cassara AM, Neufeld E, Kuster N, Tsai LH, Pascual-Leone A, Boyden ES. Noninvasive Deep Brain Stimulation via Temporally Interfering Electric Fields. Cell. 2017 Jun 1;169(6):1029-1041.e16. doi: 10.1016/j.cell.2017.05.024. PMID 28575667
- See also: Lab website for study. The Cognitive Control Lab aims to understand the neural mechanisms of goal-directed behavior, using a combination of fMRI, computational neural modeling, and neurostimulation methods in healthy and clinical human populations. — https://ccsrv1.psych.indiana.edu/cclab/
- See also: Project details for the NIMH-funded study on temporal interference stimulation, including abstract, funding, and key personnel. — https://reporter.nih.gov/project-details/11119339

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT07215299/Prot_SAP_000.pdf
  • Informed Consent Form: Informed Consent Statement Aim 1 (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT07215299/ICF_001.pdf
  • Informed Consent Form: Informed Consent Statement Aim 2 (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT07215299/ICF_002.pdf